CLINICAL TRIAL: NCT02168062
Title: A Multidisciplinary Team-Based Approach to Mitigate the Impact of Androgen Deprivation Therapy in Prostate Cancer: A Randomized Phase 2
Brief Title: Supportive Therapy in Androgen Deprivation Clinic in Improving Health Outcomes and Managing Side Effects in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 135513; NCI-2015-01058 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-05-15; First posted 2014-06-20 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Counseling; Early Intervention, Educational; Educational Status; Methods; Goserelin; Leuprolide; luprolide acetate gel depot; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): Patients receive leuprolide acetate SC or IM, goserelin acetate SC, or triptorelin pamoate IM and visit their health care provider every 3 months for 12 months. Patients will be referred to a nutrition, exercise, and symptom management service upon patient request or if deemed necessary by a healthcare provider. Patients may cross-over to Arm II after 12 months.
  Interventions: Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Drug: Triptorelin Pamoate
- Arm II (STAND clinic) (Experimental): Patients receive leuprolide acetate SC or IM, goserelin acetate SC, or triptorelin pamoate IM every 3 months for 12 months. Patients also review educational modules discussing various aspects of anti-androgen therapy and management of side effects and meet one-to-one with a licensed exercise trainer, registered dietician, and symptom management service to receive individualized counseling monthly for 12 months.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Counseling; Other: Educational Intervention; Behavioral: Exercise Intervention; Drug: Goserelin Acetate; Other: Laboratory Biomarker Analysis; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Drug: Triptorelin Pamoate

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Receive individualized nutrition counseling
  Arms: Arm II (STAND clinic)
Other: Counseling — Receive individualized symptom management service counseling
  Other Names: Counseling Intervention
  Arms: Arm II (STAND clinic)
Other: Educational Intervention — Review educational modules
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (STAND clinic)
Behavioral: Exercise Intervention — Receive individualized exercise counseling
  Arms: Arm II (STAND clinic)
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leuprolide Acetate — Given SC or IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Triptorelin Pamoate — Given IM
  Other Names: Diphereline; Pamorelin; Trelstar

SUMMARY:
This pilot partially-randomized phase II trial studies how well Supportive Therapy in Androgen Deprivation (STAND) clinic works in improving health outcomes and managing side effects in patients with prostate cancer. Individualized counseling regarding exercise and dietary habits may help improve patient understanding, satisfaction, and overall lessen adverse impact on quality of life caused by androgen deprivation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the mean percent change from baseline to 12 months in percentage body fat mass among men with prostate cancer receiving androgen deprivation therapy randomized to participate in the ?STAND? clinic versus (vs.) usual standard of care. (Randomized Cohort) II. To determine the feasibility of completing multi-disciplinary STAND clinic visits within context of concurrent chemohormonal therapy for prostate cancer. (Non-randomized Pilot Cohort)

SECONDARY OBJECTIVES:

I. To compare the mean percent change from baseline to 12 months and patterns of change over time during participation in the STAND clinic vs. usual standard of care with respect to: metabolic impact on diabetes and cardiovascular risk factors, bone health, and quality of life/psychosocial impact.

II. Among men randomized to receive usual standard of care that cross-over to participate in the STAND clinic after month 12 of the study: to measure the mean change from baseline at start of participation in the STAND clinic after 12 months of participation in: metabolic parameters including percentage body fat, fasting insulin/glucose, homeostatic model assessment insulin resistance (HOMA-IR), body weight/body mass index, waist circumference; bone health; quality of life; and patient satisfaction.

III. Among men in the non-randomized pilot cohort: to determine the mean change from baseline to 12 months during STAND clinic participation in the primary and secondary metabolic and quality of life parameters listed above.

TERTIARY OBJECTIVES:

I. To investigate for a relationship between inherited genetic polymorphisms of functional relevance near or within genes encoding proteins with roles in steroid hormone transport and androgen receptor signaling with changes in metabolic parameters among men treated with androgen deprivation therapy.

II. To investigate changes in trabecular bone micro-architecture as measured by high resolution peripheral quantitative computed tomography (QCT) Imaging of radius and tibia during androgen deprivation therapy.

III. To investigate for relationship between 2nd digit to 4th digit length ratio (2D:4D ratio) and quality of life on androgen deprivation therapy.

IV. To investigate for a relationship between 2nd digit to 4th digit length ratio and baseline empathy score as measured by validated questionnaire.

OUTLINE: Patients receiving androgen deprivation therapy are randomized to 1 of 2 arms and patients receiving concurrent chemohormonal therapy are assigned to Arm II.

ARM I (STANDARD OF CARE): Patients receive leuprolide acetate subcutaneously (SC) or intramuscularly (IM), goserelin acetate SC, or triptorelin pamoate IM and visit their health care provider every 3 months for 12 months. Patients will be referred to a nutrition, exercise, and symptom management service upon patient request or if deemed necessary by a healthcare provider. Patients may cross-over to Arm II after 12 months.

ARM II (STAND CLINIC): Patients receive leuprolide acetate SC or IM, goserelin acetate SC, or triptorelin pamoate IM every 3 months for 12 months. Patients also review educational modules discussing various aspects of anti-androgen therapy and management of side effects and meet one-to-one with a licensed exercise trainer, registered dietician, and symptom management service to receive individualized counseling monthly for 12 months.

After completion of study treatment, patients are followed up at 2, 4, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate
* Receiving or planning to receive androgen deprivation therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonist or antagonist
* Expected duration of ADT at least 12 months from date of study consent
* Concurrent antiandrogen therapy allowed but not required
* First dose of LHRH agonist or antagonist no more than 6 months prior to date of study content
* Prior/concurrent radiation allowed
* Other investigational agents in addition to LHRH agonist/antagonist are allowed (e.g. novel anti-androgens, androgen synthesis inhibitors)
* Prior androgen deprivation therapy allowed, provided there is documented evidence of testosterone recovery to > 150 ng/dL and greater than 12 months duration between last ?effective? date of ADT and date of study consent
* Randomized cohort only:

  * No prior chemotherapy within 12 months of start date of study
  * No planned chemotherapy at least 12 months from study entry
* Non-randomized pilot cohort:

  * Concurrent chemotherapy (initiated within 3 months of study entry) or planned chemotherapy within 3 months of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ? 2
* Ability to sign written informed consent
* Willing to attend monthly clinic visits at University of California, San Francisco (UCSF)

Exclusion Criteria:

* Physically unable or unwilling to participate in recommended exercise programs or travel to UCSF on a monthly basis
* Presence of permanent pacemaker or implantable medical device

  * Artificial joint prostheses and venous filters are allowed

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a small, non-randomized pilot cohort of 8 patients receiving concurrent chemohormonal therapy who were enrolled in parallel to assess the feasibility of STAND clinic participation in this patient population but were not included in the final group comparisons.
Groups:
- Arm I (Standard of Care): Patients receive leuprolide acetate subcutaneous (SC) or intramuscular (IM), or goserelin acetate SC, and visit their health care provider every 3 months for 12 months. Patients will be referred to a nutrition, exercise, and symptom management service upon patient request or if deemed necessary by a healthcare provider. Patients may cross-over to Arm II after 12 months.
  Goserelin Acetate: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Leuprolide Acetate: Given SC or IM
  Quality-of-Life Assessment: Ancillary studies
- Arm II (STAND Clinic): Patients receive leuprolide acetate SC or IM, or goserelin acetate SC every 3 months for 12 months. Patients also review educational modules discussing various aspects of anti-androgen therapy and management of side effects and meet one-to-one with a licensed exercise trainer, registered dietitian, and symptom management service to receive individualized counseling monthly for 12 months.
  Behavioral Dietary Intervention: Receive individualized nutrition counseling
  Counseling: Receive individualized symptom management service counseling
  Educational Intervention: Review educational modules
  Exercise Intervention: Receive individualized exercise counseling
  Goserelin Acetate: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Leuprolide Acetate: Given SC or IM
  Quality-of-Life Assessment: Ancillary studies
- Non-Randomized Pilot Cohort: A non-randomized pilot cohort receiving concurrent chemohormonal therapy will be enrolled in parallel to assess the feasibility of STAND clinic participation in this patient population.
Period: Overall Study
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic) | Non-Randomized Pilot Cohort
Started | 23 | 26 | 8
Completed | 23 | 26 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Randomized Pilot Cohort: A non-randomized pilot cohort of 20 patients receiving concurrent chemohormonal therapy will be enrolled in parallel to assess the feasibility of STAND clinic participation in this patient population.
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic) | Non-Randomized Pilot Cohort | Total
Number analyzed (Participants) | 23 | 26 | 8 | 57
Age, Customized [Number; unit: participants]
  50-60 years old | 4 | 7 | 3 | 14
  61-70 years old | 9 | 11 | 4 | 24
  71-80 years old | 8 | 7 | 1 | 16
  81-90 years old | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 23 | 26 | 8 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 20 | 22 | 6 | 48
  Unknown or Not Reported | 3 | 3 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 2 | 6
  White | 13 | 21 | 4 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 8 | 57

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percentage Body Fat Mass as Measured by Bioelectrical Impedance Analyzer (Randomized Cohort)
Description: The absolute change from baseline in percentage body fat after 12 months of study participation for participants in the randomized cohort was measured using a bioelectrical impedance analyzer and between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: percentage of body fat mass
Groups:
- Arm I (Standard of Care): Patients receive leuprolide acetate SC or IM, or goserelin acetate SC, and visit their health care provider every 3 months for 12 months. Patients will be referred to a nutrition, exercise, and symptom management service upon patient request or if deemed necessary by a healthcare provider. Patients may cross-over to Arm II after 12 months.
  Goserelin Acetate: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Leuprolide Acetate: Given SC or IM
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
percentage of body fat mass | -1 [-28.5 to 11.6] | 6.8 [-20.2 to 17.4]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Test type: Other; p = 0.109, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Percentage of Participants in the Non-randomized, Pilot, Cohort Who Completed Clinic Visits
Description: The percentage of participants in the pilot, non-randomized cohort who completed clinic visits for Supportive Therapy in Androgen Deprivation (STAND) will be reported to assess feasibility.
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Non-Randomized Pilot Cohort
Number analyzed (Participants) | 8
percentage of participants | 62.5

3. Secondary Outcome: Absolute Change in Blood Pressure (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in systolic and diastolic blood pressure from the baseline to month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: mmHg
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
mmHg
  Systolic Blood Pressure | 10 [-11 to 46] | 9 [-25 to 27]
  Diastolic Blood Pressure | 2 [-10 to 37] | -3 [-16 to 13]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Systolic Blood Pressure measurement comparison; Test type: Other; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Diastolic Blood Pressure measurement comparison; Test type: Other; p = 0.10, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Absolute Change in Body Weight (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in body weight from the baseline to month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: kilograms
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
kilograms | 0.8 [-8.4 to 15] | 2.6 [-11.3 to 16.8]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Weight measurement comparison; Test type: Other; p = 0.70, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Absolute Change in Percentage of Body Fat (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in percentage of body fat from the baseline to the month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: percentage of body fat
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
percentage of body fat | -1 [-28.5 to 11.6] | 6.8 [-20.2 to 17.4]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Percentage body fat measurement comparison; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Absolute Change in Waist Circumference (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in waist circumference from the baseline to the month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: centimeters
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
centimeters | 5 [-8 to 14] | 1.7 [-4 to 9.3]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Waist measurement comparison; Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Absolute Change in Hemoglobin A1c (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in percentage hemoglobin A1c from the baseline to the month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: percentage
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
percentage | -0.1 [-0.8 to 0.7] | -0.1 [-0.8 to 0.2]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Hemoglobin A1C measurement comparison; Test type: Other; p = 0.70, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Absolute Change in Insulin Resistance Score (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in insulin resistance scores from the baseline to the month 12 assessment. Insulin resistance scores were calculated using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). This calculation marks for both the presence and extent of any insulin resistance that participants might currently express. The HOMA-IR is an assessment using insulin and glucose lab values to generate an insulin resistance score. A healthy score range is 1.0 (0.5-1.4). A score of less than 1.0 means you are insulin-sensitive which is optimal. A score above 1.9 indicates early insulin resistance. A score above 2.9 indicates significant insulin resistance. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale | 0 [-1.5 to 5.4] | -0.5 [-3.1 to 3.6]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Insulin resistance score comparison; Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Absolute Change in Fasting Lipids (Randomized Cohort)
Description: Metabolic and cardiac impact for participants in the randomized cohort was measured by calculating the absolute change in fasting lipids which includes total cholesterol, low density lipoprotein, High density lipoprotein, and triglycerides levels from the baseline to the month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
milligram per deciliter (mg/dL)
  Total Cholesterol | 4 [-313 to 134] | -1 [-102 to 138]
  Low density lipoprotein | -4 [-26 to 86] | -4 [-64 to 50]
  High density lipoprotein | 5 [-18 to 46] | 7 [-70.4 to 21]
  Triglycerides | 19 [-79 to 188] | -3 [-135 to 182]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Total Cholesterol measurement comparison; Test type: Other; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Total low density lipid measurement comparison; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Total high density lipid measurement comparison; Test type: Other; p = 0.40, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Total triglyceride measurement comparison; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Absolute Change in Hours Per Week of Physical Activity Category as Measured by the Exercise Pattern Assessment (Randomized Cohort)
Description: Metabolic impact for participants from baseline to 12 months was measured using an exercise pattern questionnaire. The questionnaire measured self-reported average total time per week over the past year the participant participated in various physical activities such as walking, tennis, yoga, swimming, etc. Twelve response options for each activity are as follows: None, 1-4 minutes (min), 5-19 min, 20-39 min, 40-89 min, 1.5 hours, 2-3 hours, 4-6 hours, 7-10 hours, 11-20 hours, 21-30 hours, 31-40 hours, 40+ hours. The amount of time per week spent on each activity was converted to a hourly scale and the absolute change between baseline and month 12 times were calculated for each participant. The median absolute change in hours per week were compared for each of the 6 activity categories: non-vigorous, moderate, moderate-vigorous, vigorous, and total physical activity and total moderate and vigorous activity combined.
Time Frame: Up to 12 months
Population: Only a small subset of patients reported both baseline and 12 month data.
Measure: Median (Full Range); unit: hours per week
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 15 | 12
hours per week
  Non-vigorous physical activity | -0.62 [-10.00 to 6.54] | -1.03 [-7.30 to 2.30]
  Moderate physical activity | 0.00 [-7.00 to 7.00] | 0.00 [-8.50 to 2.50]
  Vigorous physical activity | -0.20 [-26.22 to 37.46] | -0.02 [-5.00 to 2.96]
  Total physical activity | -.30 [-19.68 to 39.26] | -.90 [-6.58 to 2.30]
  Total Moderate-Vigorous physical activity (MVPA) | -0.30 [-19.22 to 39.46] | -0.08 [-5.54 to 2.50]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Non-vigorous physical activity comparison; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Moderate physical activity comparison; Test type: Other; p = 0.979, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Moderate-Vigorous physical activity comparison; Test type: Other; p = 0.884, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Vigorous physical activity comparison; Test type: Other; p = 0.678, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Total physical activity comparison; Test type: Other; p = 0.464, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Absolute Change in Average Moderate to Vigorous Physical Activity (MVPA) as Measured by an Ambulatory Accelerometer Assessment (Randomized Cohort)
Description: Metabolic impact for participants in each group from baseline to 12 months was measured by using an ambulatory accelerometer worn by participants around their waist for 7 consecutive days. Participants were required at least 3 days of valid wear time, defined as >= 10 hours of wear per day. The accelerometer measured movement intensity and recorded vertical acceleration as "counts," providing an indication of the intensity of physical activity associated with locomotion. Non-wear time was identified using Troiano 2007 default settings in the ActiLife v6.13.3 software. The amount of time participants were engaged in moderate to vigorous physical activities (MVPA) was measured by accelerometer as counts per minute (moderate activity = 2020-5998 counts per minute, and vigorous activity = 5999 or more counts per minute). Counts are then transformed into minutes per day with a total range of 0-1440 minutes. The median absolute change in average MVPA was compared between the two groups.
Time Frame: Up to 12 months
Population: Only a small subset of patients reported both baseline and 12 month data.
Measure: Median (Full Range); unit: minutes per day
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 3 | 8
minutes per day | -18.40 [-45.46 to 39.50] | -2.36 [-26.30 to 5.90]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Average MVPA Minutes per Day Comparison; Test type: Other; p = 0.838, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Absolute Change in Bone Density T-score (Randomized Cohort)
Description: The absolute change in bone density t-scores from the baseline to the month 12 assessment for participants in the randomized cohort was measured using bone density at the lumbar spine, bone density at the femoral neck, and bone density at the total hip. A T-score of -1.0 or above is normal bone density. A T-score between -1.0 and -2.5 indicates low bone density or osteopenia. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: t-score
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
t-score
  Bone density at the lumbar spine | -2.0 [-3.50 to 0.10] | -0.40 [-1.80 to 0.60]
  Bone density at the femoral neck | -0.25 [-2.30 to 1.90] | -0.20 [-2.10 to 1.20]
  Bone density of total hip | -0.20 [-2.30 to 0.10] | -0.10 [-0.70 to 0]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Bone Density at the lumbar spine comparison; Test type: Other; p = 0.677, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Bone Density at the femoral neck comparison; Test type: Other; p = 0.493, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Bone Density of the total hip comparison; Test type: Other; p = 0.807, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Absolute Change in Serum 25-(OH) Vitamin D (Randomized Cohort)
Description: The absolute change in bone health parameters as measured by the serum 25-(OH) vitamin D level from the baseline to the month 12 assessment. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
nanograms per milliliter (ng/mL) | 3.60 [-14 to 24] | 8.10 [-21 to 20]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Serum 25-(OH) vitamin D level comparison; Test type: Other; p = 0.403, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Absolute Change in Patient Health Questionnaire-9 (PHQ-9) Scores (Randomized Cohort)
Description: The absolute change in scores on the Patient Health Questionnaire-9 (PHQ-9) from baseline after 12 months of study participation for participants was used to measure depression symptoms with a higher number indicating a greater percentage of change in scores. The total Patient Health Questionnaire-9 (PHQ-9) score is calculated by combining the responses of the participant on questions addressing how bothered the participant has been by various problems over the past 2 weeks. Each of the 9 items is scored on a scale of 0 ("Not bothered at all") to 4 ("Nearly every day"). A total score of 5-9='Mild Depression Symptoms", 10-4="Minor Depression, Major Depression (mild), or Dysthymia", 15-19="Major Depression, moderately severe", and >20="Major Depression".
  Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale | 0 [-5.0 to 3.00] | .50 [-5.0 to 3.0]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Test type: Other; p = .385, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Absolute Change in Attention Function Index (AFI) Scores (Randomized Cohort)
Description: The AFI measures a participants perceived effectiveness in functioning at time of assessment. Each of the 16 items consists of a 100 mm horizontal line anchored with opposite phrases from not at all (0 mm) to extremely well or a great deal (100 mm). Subjects are asked to place a mark on the line that best describes functioning in relation to specific activity. Scores for each item are determined by measuring distance from lower end of scale in millimeters. The total score on the instrument is computed by obtaining an average of 16 scales. The absolute change in score by group from baseline up to month 12 in Attention Function Index was used to measure perceived effectiveness in common activities requiring attention and working memory in daily life with a higher number indicating a greater absolute change in scores. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Population: Only a subset of patients reported both baseline and 12 month data.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 15 | 11
score on a scale | 2.31 [-27.75 to 26.62] | -4 [-15.26 to 10.44]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Attention Function Index (AFI) Score Comparison; Test type: Other; p = .148, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Absolute Change in the 12-item Short Form Survey (SF-12) Assessment Item Scores for Patients in the Randomized Cohort
Description: The SF-12 is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. The SF-12 consists of a subset of 12 items from the SF-36® Health Survey (SF-36) and measures two composite outcomes assessing mental health composite score (MCS) and physical health composite scores (PCS). The PCS & MCS are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The absolute change in item score by group from baseline up to 12 months was used to assess the quality of life/psychosocial impact on the patients with a larger scores indicating a greater degree of change on physical and mental health. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Population: Only a subset of participants completed questionnaires at both baseline and 12 months.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 20 | 25
score on a scale
  Mental Composite Score | 4.81 [-8.46 to 11.90] | -2.37 [-7.37 to 4.03]
  Physical Composite Score | -2.90 [-17.82 to 18.75] | -1.60 [-6.65 to 8.59]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Mental Composite Score Comparison; Test type: Other; p = .077, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Physical Composite Score Comparison; Test type: Other; p = 0.401, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Absolute Change in International Prostate Symptom Score (IPSS) (Randomized Cohort)
Description: The absolute change in score by group from baseline up to month 12 on the International Prostate Symptom Score (IPSS) was used to measure the severity of lower urinary tract symptoms and erectile function with lower numbers indicating less change in symptoms. Seven questions with scores ranging from 1-5 are summed to create a total score. Scores of 1-7 indicate mild symptoms, scores of 8-19 indicate moderate symptoms, and scores of 20-35 indicate severe symptoms. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale | 2 [-20 to 24] | -2 [-9 to 22]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Test type: Other; p = 0.085, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Absolute Change in Last Question on International Prostate Symptom Score (IPSS) (Randomized Cohort)
Description: The absolute change in score by group from baseline up to month 12 on the International Prostate Symptom Score (IPSS) was used to measure the severity of lower urinary tract symptoms and erectile function. The last question on the IPSS can be looked at separately from the total score as it asks the participants to rate the overall quality of life due to their existing urinary symptoms on a scale of 0-6, with lower scores indicating a better quality of life. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale | 0 [-3 to 2] | 0 [-1 to 1]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Test type: Other; p = 0.676, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Absolute Change in Hot Flash Related Daily Interference Scale Score (HFRDIS) (Randomized Cohort)
Description: The absolute change in Hot Flash Related Daily Interference Scale from baseline to month 12 was used to measure the impact of occurrence of hot flashes on daily activities with higher numbers indicating a greater change in the interference of hot flashes with participant's quality of life. The HFRDIS is a 10-item scale measuring the degree hot flashes interfere with nine daily activities; the tenth item measures the degree hot flashes interfere with overall quality of life. The HFRDIS was developed to include daily life activities specific to impact of hot flashes. Participants rate degree to which hot flashes have interfered with each item during previous week using a 0 (do not interfere) to 10 (completely interfere) point scale, with total score ranging from 0-100. Higher scores indicate higher interference and thus, greater impact on quality of life. Women without hot flashes are asked to mark 0 for each item. Group comparisons performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale | 13 [-22 to 67] | 4.5 [-52 to 37]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Test type: Other; p = 0.183, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Absolute Change in Expanded Prostate Cancer Index Composite Short Form (EPIC-26) Scores to Assess Erectile and Urinary Function (Randomized Cohort)
Description: The EPIC-26 was measured at baseline and month 12 to determine the impact of quality of life issues across 5 prostate cancer specific domains: Urinary incontinence, Urinary irritation, Bowel function, Sexual function, and Hormonal function and overall total quality of life. Response options for each EPIC item form a Likert scale, and the raw score of each item is then transformed linearly to a 0-100 scale. Multiple items are combined and then averaged to form the domain scores and total score at each time point also ranging from 0-100, with higher scores representing better health related quality of life (HRQOL). Between group comparisons were performed using the Wilcoxon-rank-sum test
Time Frame: Up to 12 months
Population: Only a subset of patients reported both baseline and 12 month data.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 25 | 20
score on a scale
  Total | -4.91 [-25.53 to 17.10] | -3.85 [-11.54 to 11.27]
  Urinary incontinence | 0 [-37.75 to 39.50] | 0 [-20.57 to 17.00]
  Urinary irritation | -5.00 [-27.50 to 60.00] | 5.00 [-5.00 to 25.00]
  Bowel function | 0 [-87.50 to 25.00] | -4.17 [-16.67 to 12.50]
  Sexual function | -12.50 [-47.00 to 16.67] | -2.08 [-48.67 to 12.50]
  Hormonal Function | 0 [-41.25 to 12.50] | -17.50 [-35.00 to 25.00]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Total Score Comparison; Test type: Other; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Urinary Incontinence Score Comparison; Test type: Other; p = 0.844, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Urinary Irriation Score Comparison; Test type: Other; p = 0.175, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Bowel Function Score Comparison; Test type: Other; p = 0.472, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Sexual Function Score Comparison; Test type: Other; p = 0.405, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); EPIC-26 Hormonal Function Score Comparison; Test type: Other; p = 0.749, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Absolute Change in Lee Fatigue Scale Scores (Randomized Cohort)
Description: The absolute change in Lee Fatigue Scale from baseline to month 12 was used to measure the impact of Fatigue on a participants quality of life. The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X" representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired"). Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10). The fatigue subscale score is calculated as the mean of the 13 fatigue items, and the energy subscale score is the mean of the 5 energy items. Higher scores on the fatigue subscale represent greater fatigue severity, and higher scores on the energy subscale indicate higher levels of energy. Between group comparisons were performed using the Wilcoxon-rank-sum test.
Time Frame: Up to 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic)
Number analyzed (Participants) | 23 | 26
score on a scale
  Fatigue Scale | 5.68 [-36.09 to 33.38] | 3.15 [-5.40 to 29.15]
  Energy Scale | -0.10 [-19.80 to 44.20] | 1.30 [-15.60 to 27.40]
Statistical Analysis 1: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Fatigue Scale Score Comparison; Test type: Other; p = 0.907, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Standard of Care) vs Arm II (STAND Clinic); Energy Scale Score Comparison; Test type: Other; p = 0.792, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The Behavioral-Dietary intervention under investigation was not determined to pose any significant risk to the patient however, all grade(s) 3-5 adverse events, whether or not unexpected, and whether or not considered to be associated with the use of the study treatment were collected.
Arm/Group | Arm I (Standard of Care) | Arm II (STAND Clinic) | Non-Randomized Pilot Cohort
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26 | 0/8
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26 | 0/8

LIMITATIONS AND CAVEATS:
Absolute change calculated for outcomes and and non-parametric statistical tests performed due to small sample size from early study termination. Non-randomized pilot cohort to assess feasibility was not included in group comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT02168062/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT02168062/ICF_001.pdf